CLINICAL TRIAL: NCT03547999
Title: A Phase II Trial of Perioperative CV301 Vaccination in Combination With Nivolumab and Systemic Chemotherapy for Resectable Hepatic-Limited Metastatic Colorectal Cancer HCRN: GI16-288
Brief Title: A Trial of Perioperative CV301 Vaccination in Combination With Nivolumab and Systemic Chemotherapy for Metastatic CRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drugs Unavailable
Sponsor: Patrick Boland (Other)
Collaborators: Bavarian Nordic (Industry); Hoosier Cancer Research Network (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Patrick Boland, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GI16-288
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: CV301 Vaccination; mFOLFOX6; Fowlpox (FP)-CV301; nivolumab; MVA-BN-CV301
MeSH Terms: conditions — Colorectal Neoplasms; Fowlpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic; Nivolumab

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A - Control (Active Comparator): mFOLFOX6 and Nivolumab every 2 weeks for 4 cycles. After neoadjuvant therapy, patients will be re-evaluated for surgical resection. Patients still considered resectable will undergo surgical resection with the goal of completely treating all of their disease by either resection and/or ablation. Patients with bilobar disease must have all of their disease treated in a single operation. Once patients in the post-operative period are deemed ready to begin therapy, patients in the control arm will then undergo another 8 cycles of mFOLFOX6 in addition to Nivolumab. After this, Nivolumab will be given every 4 weeks completing therapy at week 110.
  Interventions: Drug: mFOLFOX6; Drug: Nivolumab
- Arm B - Experimental (Experimental): Two doses of Nivolumab and MVA-BN-CV301 each given 2 weeks apart (Days -28, -14), followed by four doses of Nivolumab plus FPV-CV301 given 2 weeks apart concurrently with mFOLFOX6, which will again be administered every 2 weeks for 4 cycles (Nivolumab, FPV-CV301 and mFOLFOX6). After neoadjuvant therapy, patients will be re-evaluated for surgical resection. Patients still considered resectable will undergo surgical resection with the goal of completely treating all of their disease by either resection and/or ablation. Patients with bilobar disease must have all of their disease treated in a single operation. Patients in the experimental arm will receive 8 cycles of mFOLFOX6 in addition to Nivolumab and FVP-CV301 boosters with the first two given on Day 0 and 14 and then every 4 weeks. FVP-CV301 will then be administered every twelve weeks completing therapy at week 110.
  Interventions: Drug: mFOLFOX6; Biological: MVA-BN-CV301; Biological: FPV-CV301; Drug: Nivolumab

INTERVENTIONS:
Drug: mFOLFOX6 — The control arm (Arm A) and experimental arm (Arm B) will receive mFOLFOX6 every 2 weeks for 4 cycles. Once patients in the post-operative period are deemed ready to begin therapy, patients in the control arm will then undergo another 8 cycles of mFOLFOX6.
Biological: MVA-BN-CV301 — The experimental arm (Arm B) will receive MVA-BN-CV301 in 4 injections of 4 x 10(8) infectious units/0.5 mL given subcutaneously prior to the start of chemotherapy on days -28 and -14.
  Other Names: Modified Vaccinia Ankara; CV301
  Arms: Arm B - Experimental
Biological: FPV-CV301 — The experimental arm (Arm B) will receive FPV-CV301 in 1 dose of 1 x 10(9) infectious units/0.5 mL given subcutaneously concurrently with chemotherapy (at least an hour prior to chemotherapy) on days 0, 14, 28 and 42 pre-operatively, and FVP-CV301 boosters on day 0 and 14 and then every 4 weeks (day 42, 70, 98). After day 98, FVP-CV301 will then be administered every twelve weeks completing therapy at week 110.
  Other Names: Fowl Pox Virus
  Arms: Arm B - Experimental
Drug: Nivolumab — Nivolumab at a dose of 240 mg as a 30 minute IV infusion every 2 weeks until progression. Arm B will receive Nivolumab starting with the vaccinations. Arm A will begin the Nivolumab with the initiation mFOLFOX.
  Other Names: Opdivo

SUMMARY:
This is a multi-center Phase II randomized study. We plan to enroll 78 patients with biopsy-proven hepatic-limited metastatic colorectal cancer deemed resectable after multi-disciplinary discussion. Eligible patients must have confirmed isolated liver metastases by radiographic imaging of the investigators' choosing. Imaging must include the chest, abdomen, and pelvis regardless of imaging modality chosen. Patients will be randomized to either the control arm or the experimental arm. The control arm will receive mFOLFOX6 every 2 weeks for 4 cycles concurrently with Nivolumab. The experimental arm will first be treated with 2 vaccinations of MVA-BN-CV301 given two weeks apart (Days -28, -14) concurrently with Nivolumab followed by 4 vaccinations of FPV-CV301 given two weeks apart concurrently with mFOLFOX6 and Nivolumab, which will again be administered every 2 weeks for 4 cycles (FPV-CV301, mFOLFOX6 and Nivolumab) After Cycle 4, patients will be re-evaluated for surgical resection by re-staging CT chest, abdomen and pelvis (C/A/P). Patients still considered resectable will undergo surgical resection with the goal of complete resection. Patients who cannot be completely resected will continue to be followed on study, and an additional appropriate candidate will be randomized to the corresponding arm.

We will collect peripheral blood and tumor tissue at the time of surgical resection, if applicable, or by re-biopsy if resection is not possible. Post-operative therapy will begin when patients are deemed ready by their surgical oncologist team. Patients in the control arm will then undergo another 8 cycles of mFOLFOX6 with Nivolumab administered concurrently. Nivolumab will then be administered every four weeks. The experimental arm will receive the same post-operative regimen but including FPV-CV301 boosters given concurrently with mFOLFOX6 and Nivolumab. FPV-CV301 will then be administered every 12 weeks, and Nivolumab every 4 weeks. We will collect peripheral blood for evaluation of correlates upon the completion of therapy. The vaccination approach of initial immunization during the neoadjuvant period followed by FPV-CV301 boosters for two years postoperatively was chosen to optimize the induction of a long-lasting tumor-specific host response. Neoadjuvant vaccination will also allow for analysis of the tumor microenvironment in resection specimens.

Post-therapy patients will be under surveillance per NCCN guidelines with repeat CEA every 3 months for 2 years followed by every 6 months for 1 year (total 3 years), repeat CT of the C/A/P every 3 months for 2 years followed by every 6 months for up to 1 year (total 3 years), and colonoscopy at one year with repetition based on findings at the time of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 2 and/or sufficient to undergo both perioperative systemic chemotherapy and hepatic surgery as determined by surgical and medical oncology evaluations.
* Histologically confirmed hepatic-limited metastatic colorectal cancer.
* Genomic testing results are required. FoundationOne platform is preferred, however results from an equivalent genomic platform may be used after discussion with the sponsor investigator.
* Completely resectable disease as determined by the guidelines below and surgical oncology evaluation. Patients with bilobar disease that requires resection and ablation are allowed provided the surgical oncologist can render the patient NED (no evidence of disease) at the conclusion of the operation. Synchronous primary colorectal and metastatic hepatic tumors are eligible, provided all disease can be resected in a single operation. NOTE: Subjects who had surgery for their primary tumor prior to registration to this trial are still eligible. Additionally:

  * No radiographic evidence of involvement of: extrahepatic bile ducts, main portal vein or celiac/retroperitoneal lymph nodes.
  * Adequate predicted functional liver remnant (FLR) as deemed by the individual site surgical oncologists.
* Patients with synchronous metastatic disease are allowed provided their primary tumor can be completely resected at the time of metastasectomy. Neoadjuvant pelvic radiotherapy for rectal cancer is not permitted
* Patients must be treatment naïve with respect to their stage IV colorectal cancer. History of prior adjuvant systemic chemotherapy containing oxaliplatin is allowed as long as as it has been greater than 12 months from completion of oxaliplatin to study enrollment. NOTE: Neoadjuvant pelvic chemoradiotherapy as part of the management of synchronous metastatic rectal cancer is allowed, provided chemoradiation was completed prior to enrollment on study.
* Hematological:

  * Platelet Count ≥ 100,000 mm^3
  * Absolute Neutrophil Count (ANC) ≥1500 µ/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
* Renal:

  o Creatinine < 1.5 x ULN OR Calculated Creatinine Clearance ≥ 60 mL/min
* Hepatic:

  * Total Bilirubin ≤ 1.5 × upper limit of normal (ULN)^2
  * Aspartate aminotransferase (AST) ≤ 5 × ULN; given presence of liver metastases
  * Alanine aminotransferase (ALT) ≤ 5 × ULN; given presence of liver metastases
  * Alkaline Phosphatase < 2.5 x ULN
  * INR, PT, or APTT ≤ 1.5x ULN unless participant is receiving anticoagulant therapy, in which case they must be on a stable dose
* Females of childbearing potential must have a negative serum pregnancy test within 24 hours of study drug. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months without another cause, or a documented serum follicle stimulating hormone (FSH) ≥ 35 mIU/mL. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Females of childbearing potential and male participants must be willing to abstain from heterosexual intercourse or to use contraception as outlined in the protocol.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Patients with mutations in or deficient expression of one or more of the mismatch repair genes listed: MSH2, MSH3, MSH6, MLH1, PMS1, PMS2.
* Active infection requiring systemic therapy.
* Pregnant or breastfeeding.
* Second primary malignancy. Clear exceptions are 1) patient had a second primary malignancy but has been treated and disease free for at least 3 years and, 2) in situ carcinoma (e.g. in situ carcinoma of the cervix). Patients with chronic lymphocytic leukemia will be allowed if their blood counts are within acceptable hematologic parameters and if they are not currently requiring cytotoxic or biologic anticancer treatment (supportive treatment such as IVIG is permitted).
* Metastatic disease not limited to the liver.
* Disease not amenable to complete resection, not resectable within the confines of a single surgery, or where resection would result in inadequate functional liver remnant.
* Prior surgery or systemic therapy for colorectal cancer within 6 months or 12 months if systemic chemotherapy included oxaliplatin of study enrollment.
* Immunodeficient patients including but not limited to patients with HIV/AIDS and chronic Hepatitis B and C.
* Patient with clinically significant cardiomyopathy, coronary disease, heart failure New York Heart Association (NYHA) class III or IV, or cerebrovascular accident (CVA) within 1 year of study enrollment (CV301).
* Subjects with known severe allergy to eggs, egg products, or aminoglycoside antibiotics (for example, gentamicin or tobramycin) (CV301).
* Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Participants with history of life-threatening toxicity related to prior immune therapy (eg. anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (e.g. Hormone replacement after adrenal crisis)
* Excluding patients with serious or uncontrolled medical disorders
* Treatment with botanical preparations (e.g. herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to randomization/treatment.
* History of allergy or hypersensitivity to study drug components.
* History of allogenic stem cell or solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boland, M.D., Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center Research Institute, Inc., Westwood, Kansas
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — https://hoosiercancer.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Control: mFOLFOX6 and Nivolumab every 2 weeks for 4 cycles. After neoadjuvant therapy, patients will be re-evaluated for surgical resection. Once patients in the post-operative period are deemed ready to begin therapy, patients in the control arm will then undergo another 8 cycles of mFOLFOX6 in addition to Nivolumab. After this, Nivolumab will be given every 4 weeks completing therapy at week 110.
  mFOLFOX6: Arm A will receive mFOLFOX6 every 2 weeks for 4 cycles. Once patients in the post-operative period are deemed ready to begin therapy, patients in the control arm will then undergo another 8 cycles of mFOLFOX6.
  Nivolumab: Nivolumab at a dose of 240 mg as a 30 minute IV infusion every 2 weeks until progression. Arm B will receive Nivolumab starting with the vaccinations. Arm A will begin the Nivolumab with the initiation mFOLFOX.
- Arm B - Experimental: Two doses of Nivolumab and MVA-BN-CV301 will given 2 weeks apart (Days -28, -14), followed by four doses of Nivolumab plus FPV-CV301 given 2 weeks apart concurrently with mFOLFOX6 for 4 cycles. After neoadjuvant therapy, patients will be re-evaluated for surgical resection. Once patients in the post-operative period are deemed ready to begin therapy, patients will receive 8 cycles of mFOLFOX6 in addition to Nivolumab and FVP-CV301 boosters with the first two given on Day 0 and 14 and then every 4 weeks.
  mFOLFOX6: Arm B will receive mFOLFOX6 every 2 weeks for 4 cycles. Once patients in the post-operative period are deemed ready to begin therapy, patients will then undergo another 8 cycles of mFOLFOX6.
  MVA-BN-CV301: Arm B will receive MVA-BN-CV301 in 4 injections of 4 x 10(8) infectious units/0.5 mL given subcutaneously prior to the start of chemotherapy on days -28 and -14.
  FPV-CV301: Arm B will receive FPV-CV301 in 1 dose of 1 x 10(9) infectious units/0.5 mL given subcutaneously concurrently with chemotherapy on days 0, 14, 28 and 42 pre-operatively, and FVP-CV301 boosters on day 0 and 14 and then every 4 weeks (day 42, 70, 98). After day 98, FVP-CV301 will then be administered every twelve weeks completing therapy at week 110.
  Nivolumab: Nivolumab at a dose of 240 mg as a 30 minute IV infusion every 2 weeks until progression.
Period: Overall Study
Arm/Group | Arm A - Control | Arm B - Experimental
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Control | Arm B - Experimental | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Median (Full Range); unit: years] | 60 [51 to 71] | 61 [35 to 72] | 61 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 9 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    ECOG = 0 | 6 | 7 | 13
    ECOG = 1 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: 3-year Overall Survival (OS) Rate From Metastasectomy
Description: 3-year Overall Survival (OS) rate is defined as the percentage of patients who are still alive at 3 years.
Time Frame: 3 years
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Overall survival was defined as all patients receive one dose of protocol therapy and are completely resected.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Control | Arm B - Experimental
Number analyzed (Participants) | 7 | 9
Percentage of participants | 100 | 100

2. Secondary Outcome: 3-Year Recurrence Free Survival (RFS) Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response(CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  The 3-year recurrence-free survival (RFS) rate is defined as the percentage of patients who have not experienced disease recurrence three years after treatment, as calculated using Kaplan-Meier survival analysis.
Time Frame: 3 years
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Recurrence free survival was defined as all patients receive one dose of protocol therapy and are completely resected.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Control | Arm B - Experimental
Number analyzed (Participants) | 7 | 9
Percentage of participants | 53.6 | 61

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response(CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR = CR +PR
Time Frame: Up to 57 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoints Overall Response Rate was defined as all patients receive one dose of protocol therapy and are completely resected.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Control | Arm B - Experimental
Number analyzed (Participants) | 7 | 9
Percentage of participants | 57.14 | 100

4. Secondary Outcome: Patients Amenable to Complete Resection/Ablation
Description: Compare the percentage of patients amenable to complete resection/ablation between the experimental and control treatment groups in patients who experience a recurrence after surgery
Time Frame: Up to 57 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoints Percentage of patients amenable to complete resection/ablation was defined as all patients who experience a recurrence after surgery.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Control | Arm B - Experimental
Number analyzed (Participants) | 5 | 3
Percentage of participants | 40 | 0

5. Secondary Outcome: Perioperative Surgical Outcomes
Description: The Clavien-Dindo classification will be used for grading the severity of postoperative complications. It provides a standardized way to report and compare surgical outcomes, based on the therapy required to treat a complication. It grades from 1 to 5 where 1= Any deviation from normal postoperative course without need for pharmacological, surgical, endoscopic, or radiological interventions. Acceptable treatments: antiemetics, antipyretics, analgesics, physiotherapy, wound dressings.
  2 = Requires pharmacological treatment with drugs other than those allowed for Grade 1. Includes blood transfusions, antibiotics and total parenteral nutrition (TPN). 3 = Requiring surgical, endoscoptic or radiological intervention. 3a = Intervention under regional/local anesthesia. 3b = Intervention under general anesthesia. 4= Life-threatening complication requiring intensive care/intensive care unit management.4a= Single organ dysfunction. 4b= Multi-organ dysfunction. 5 = Patient demise.
Time Frame: Up to 6 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoints Perioperative Surgical Outcomes was defined as all patients receive one dose of protocol therapy and are completely resected.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Control | Arm B - Experimental
Number analyzed (Participants) | 7 | 9
Participants
  Grade = 1 | 4 | 4
  Grade = 2 | 1 | 2
  Grade = 3 | 0 | 1
  Grade = 3b | 2 | 2

6. Secondary Outcome: 3-Year Overall Survival (OS) Rate From Registration
Description: 3-Year OS (Overall Survival) rate is defined as the percentage of patients who are still alive at 3 years.
Time Frame: 3 years
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Control | Arm B - Experimental
Number analyzed (Participants) | 8 | 9
Percentage of participants | 100 | 100

7. Secondary Outcome: Pathologic Response Rate
Description: Compare the pathologic response rate to neoadjuvant therapy in resected tumor tissue between the experimental and control groups. Pathologic Response Rate refers to the percentage of patients whose tumors show a specific level of response after it has been surgically removed.
Time Frame: Up to 6 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoints pathologic response was defined as all patients receive one dose of protocol therapy and are completely resected.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Control | Arm B - Experimental
Number analyzed (Participants) | 7 | 9
Percentage of participants | 71.4 | 100

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Arm A - Control | Arm B - Experimental
All-Cause Mortality (participants affected / at risk) | 0/8 | 1/9
Serious Adverse Events (participants affected / at risk) | 6/8 | 5/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Control (N=8) | Arm B - Experimental (N=9)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (2)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 1 (3)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 1 (1) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 0 (0) | 1 (4)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Control (N=8) | Arm B - Experimental (N=9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 4 (6)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (13) | 7 (33)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 (6) | 6 (18)
ANEMIA (Blood and lymphatic system disorders) | 6 (12) | 6 (26)
ANOREXIA (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (10) | 7 (31)
BLOATING (Gastrointestinal disorders) | 2 (2) | 2 (3)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (9) | 1 (5)
BLURRED VISION (Eye disorders) | 1 (1) | 2 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CHILLS (General disorders) | 2 (2) | 4 (6)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 6 (6) | 2 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
CREATININE INCREASED (Investigations) | 3 (7) | 1 (3)
DIARRHEA (Gastrointestinal disorders) | 5 (6) | 8 (14)
DIZZINESS (Nervous system disorders) | 1 (1) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 2 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 1 (2) | 4 (7)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
EDEMA LIMBS (General disorders) | 2 (3) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 5 (8) | 7 (17)
FEVER (General disorders) | 3 (3) | 3 (7)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (4) | 4 (4)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (2) | 2 (3)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (3) | 3 (8)
HEMATOMA (Vascular disorders) | 1 (2) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (14) | 7 (27)
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
HYPERNATREMIA (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
HYPERTENSION (Vascular disorders) | 4 (9) | 5 (15)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 4 (9) | 4 (11)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 4 (12) | 4 (12)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 (3) | 4 (9)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 4 (5) | 4 (9)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (6) | 6 (12)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (6) | 3 (6)
HYPOTENSION (Vascular disorders) | 2 (2) | 2 (3)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 1 (1)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 1 (1) | 0 (0)
INR INCREASED (Investigations) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 4 (6)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 2 (2) | 3 (4)
LIPASE INCREASED (Investigations) | 7 (20) | 5 (26)
LYMPHOCYTE COUNT DECREASED (Investigations) | 4 (12) | 5 (20)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (4) | 3 (4)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 3 (4) | 6 (17)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 6 (13) | 7 (18)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
PAIN (General disorders) | 2 (3) | 3 (3)
PARESTHESIA (Nervous system disorders) | 1 (1) | 2 (3)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 6 (9) | 9 (21)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 6 (16) | 6 (11)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (8) | 3 (5)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
SERUM AMYLASE INCREASED (Investigations) | 7 (11) | 4 (12)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 3 (5) | 2 (7)
THROMBOEMBOLIC EVENT (Vascular disorders) | 3 (4) | 0 (0)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (2) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 4 (4) | 3 (3)
WEIGHT GAIN (Investigations) | 1 (1) | 0 (0)
WEIGHT LOSS (Investigations) | 1 (3) | 1 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 4 (10) | 5 (18)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
BLADDER SPASM (Renal and urinary disorders) | 0 (0) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 1 (1)
CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1)
CPK INCREASED (Investigations) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ERYTHRODERMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 0 (0) | 2 (2)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 2 (3)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 0 (0) | 3 (10)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HOT FLASHES (Vascular disorders) | 0 (0) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (11)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 0 (0) | 3 (5)
INJECTION SITE REACTION (General disorders) | 0 (0) | 7 (10)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
MALAISE (General disorders) | 0 (0) | 1 (1)
MUSCLE WEAKNESS TRUNK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NAIL LOSS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 1 (4)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 0 (0) | 1 (1)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03547999/Prot_SAP_000.pdf